CLINICAL TRIAL: NCT00224900
Title: Development of a Life Skills Intervention for Young Adolescents Perinatally-Infected With HIV and Their Caregivers Part A: Focus Group And Measurement Evaluation
Brief Title: Development of a Life Skills Intervention for Young Adolescents Perinatally-Infected With HIV and Their Caregivers
Status: Terminated | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 045a
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infection
Keywords: Perinatally-acquired HIV infection; Life Skills; Focus Group; Young adolescents; Caregivers
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
During this phase of the study, a focus group will be conducted with young adolescents perinatally infected with HIV and with their caregivers to develop and evaluate the content of the proposed intervention. The purpose of the focus groups is to identify key issues and challenges that often face young adolescents perinatally infected with HIV and their caregivers as well as to elicit suggestions to enhance the feasibility and acceptability of the proposed intervention. The focus groups will be audio recorded and transcribed and reviewed by all involved in future protocol development. Themes will be pulled directly from the focus groups to guide examples and areas of emphasis in the intervention. In addition, proposed measures will be administered to the adolescents and their caregivers and assessed for appropriateness for this population.

DETAILED DESCRIPTION:
This study is designed to collect information from HIV-1 perinatally infected adolescents for the development of a pilot study that will use a life skills intervention model. One focus group comprised of adolescents and one focus group comprised of their caregivers will use a series of open-ended questions to facilitate a group discussion to define the life skills intervention model. Ten young adolescents, ages 11 to 14 years, and their caregivers will participate in these focus groups at Rainbow Babies and Children's Hospital in Cleveland, Ohio. The protocol will be site-restricted for participation. The responses from the focus group will be used to tailor the proposed life skills intervention model and to provide a detailed description of intervention content including: common peer issues of young adolescents perinatally infected with HIV, typical sexual knowledge and behaviors, typical areas of conflict between adolescents and caregivers, and common ways of managing conflict. In addition, those that participate in the focus group will be asked to complete a series of questionnaires in order to assess the appropriateness of the proposed measurement battery for adolescents perinatally infected with HIV and their caregivers.

Findings from this study (ATN 045- Part A) will be used in the development of a proposal for a pilot study of the life skills intervention model (ATN 045-Part B). The pilot study will examine the feasibility of successfully providing a life skills intervention to HIV-1 infected young adolescents at an ATN clinical site, the acceptability of such an intervention in young adolescents, as well as the logistics of providing such an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinically-identified HIV-1 infected subjects 11-14 years of age and their caregivers.
* HIV status has been disclosed to the adolescent.
* HIV-1 infection transmission due to perinatal infection as identified by treating physician.
* Caregiver is legal guardian of the adolescent as indicated by the medical team in the clinic from which recruitment will be conducted.
* Adolescent lives with the caregiver.
* Adolescent and caregiver speak English.

Exclusion Criteria:

* Caregiver permission denied or adolescent does not assent.
* Adolescent previously diagnosed as mentally retarded as reported by caregiver through school and/or other psychological testing.
* Adolescent and/or caregiver too medically fragile. Medically fragile is functionally defined as being physically unable to attend the group.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young adolescents perinatally infected with HIV, 11 to 14 years of age and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahna L Hoff, Ph.D., Study Chair — Case Western Reserve University School of Medicine and Rainbow Babies and Childrens Hospital
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org